CLINICAL TRIAL: NCT02456727
Title: Acupuncture Approaches to Decrease Disparities in Outcomes of Pain Treatment - A Two Arm Comparative Effectiveness Trial
Brief Title: Acupuncture Approaches for Chronic Pain
Acronym: AADDOPT-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Montefiore Medical Center (Other); Mount Sinai Beth Israel Department of Integrated Medicine (Unknown); Pacific College of Oriental Medicine (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Diane Mckee, Prof. Family and Social Medicine, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-4192; AD-1402-10857 (Other: PCORI)
Record Dates: First submitted 2015-03-31; First posted 2015-05-28 (Estimated); Results first posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-08

CONDITIONS: Chronic Pain; Osteoarthritis; Neck Pain; Back Pain
Keywords: Acupuncture; Group/Community Acupuncture; Individual Acupuncture; Chronic Pain; Underserved; Urban Primary Care; Osteoarthritis; Back Pain; Neck Pain
MeSH Terms: conditions — Chronic Pain; Osteoarthritis; Neck Pain; Back Pain | interventions — Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual Acupuncture (Active Comparator): Participants will be treated weekly with individual acupuncture treatment sessions for 12 consecutive weeks. Quality of life assessments will be taken at intervals during treatment and post-treatment.
  Interventions: Procedure: Individual Acupuncture
- Group/Community Acupuncture (Active Comparator): Participants will be treated weekly with group acupuncture treatments sessions for 12 consecutive weeks. Quality of life assessments will be taken at intervals during treatment and post-treatment.
  Interventions: Procedure: Group/Community Acupuncture

INTERVENTIONS:
Procedure: Group/Community Acupuncture — Acupuncture treatment in a group setting.
  Arms: Group/Community Acupuncture
Procedure: Individual Acupuncture — Acupuncture treatment in an individual setting.
  Arms: Individual Acupuncture

SUMMARY:
Chronic pain is a major public health problem that places many burdens on individuals, including impairment of physical and psychological functioning, lost productivity, and side effects of medications used to treat pain. There is also substantial evidence that minority populations differ both in prevalence and outcomes of chronic pain; access to care is a key component in these differences. Strong evidence now supports the use of acupuncture in the treatment of chronic pain conditions, including when provided in the primary care setting to participants from ethnically diverse, medically underserved populations. Acupuncture is slowly being integrated into pain management in many conventional health care settings, but cost and reimbursement for this service remain obstacles to offering acupuncture, especially in primary care and safety net settings. Because group acupuncture can be offered at much lower cost, demonstrating that individual and group delivery are equally effective could reduce barriers to use of this effective pain management approach.

The primary aim of this study will be to evaluate whether acupuncture delivered in the group setting for participants with chronic pain is equal to acupuncture delivered in the individual setting. A secondary objective will be to use qualitative analysis to understand and describe the participants' experience of both acupuncture approaches, and to utilize this data to inform intervention delivery and dissemination, to better incorporate the participants' perspective.

ELIGIBILITY:
Inclusion Criteria:

* Referred by a primary care provider from one of our participating primary care health centers
* Provider-documented diagnosis of osteoarthritis (any joint), neck pain, OR back pain
* Self-reported pain score of ≥4 for at least 3 months prior to program entry
* Able to provide consent for treatment and data collection in either English or Spanish

Exclusion Criteria:

* < 21 years of age
* Chronic pain not documented OR self reported pain of ≥4 for less than 3 months.
* Currently taking oral or injectable anticoagulants.
* Lack of contact information OR unavailable for duration of entire treatment period (24 weeks)
* Inability to consent to treatment and data collection.
* Active psychosis
* Active substance abuse

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 779 (Actual)
Dates: Start 2015-05; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Diane McKee, MD, MS, Principal Investigator — Albert Einstein College of Medicine; Benjamin Kligler, MD, Principal Investigator — Mount Sinai Beth Israel
Locations (1):
- Montefiore Medical Group, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McKee MD, Nielsen A, Anderson B, Chuang E, Connolly M, Gao Q, Gil EN, Lechuga C, Kim M, Naqvi H, Kligler B. Individual vs. Group Delivery of Acupuncture Therapy for Chronic Musculoskeletal Pain in Urban Primary Care-a Randomized Trial. J Gen Intern Med. 2020 Apr;35(4):1227-1237. doi: 10.1007/s11606-019-05583-6. Epub 2020 Feb 19. PMID 32076985

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were referred by their primary care providers (PCPs) from their participating health care center. For patients who met the eligibility criteria, PCPs completed a study-specific referral form and obtained permission to contact the patient by phone. Participants were then contacted by the study staff and screened for eligibility.
Pre-assignment Details: Participants were screened by phone and completed an oral consent. They were mailed a treatment consent form and told to contact the study team in order to complete the baseline and receive their treatment arm. Several participants were excluded for various reasons including ineligibility and declining participation.
Groups:
- Group Acupuncture: Participants who were randomized to receive acupuncture weekly in a group acupuncture setting for 12 consecutive weeks.
- Individual Acupuncture: Participants who were randomized to receive acupuncture weekly in an individual acupuncture setting for 12 consecutive weeks.
Period: Overall Study
Arm/Group | Group Acupuncture | Individual Acupuncture
Started (Participants who were baselined and completed an oral consent.) | 389 | 390
Initiated Treatment (Participants who signed the treatment consent form and attended at least one session of acupuncture.) | 346 | 360
6 Week (Patients who completed the week 6 follow up questionnaires.) | 298 | 320
12 Week (Patients who completed the week 12 follow up questionnaires.) | 295 | 310
24 Week (Patients who completed the week 24 follow up questionnaires.) | 280 | 284
Completed | 280 | 284
Not Completed | 109 | 106
Not completed — Lost to Follow-up | 63 | 65
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 1 | 10
Not completed — Never Initiated Treatment | 43 | 30

BASELINE CHARACTERISTICS:
Population: All participants who were randomized to receive acupuncture weekly in either a group or an individual acupuncture setting for 12 consecutive weeks.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Acupuncture | Individual Acupuncture | Total
Number analyzed (Participants) | 389 | 390 | 779
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 316 | 303 | 619
  >=65 years | 73 | 87 | 160
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.19 (13.77) | 55.44 (13.20) | 54.80 (13.49)
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Median | 54.93 [45.87 to 62.44] | 55.42 [47.45 to 63.96] | 55.19 [46.78 to 63.20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 315 | 312 | 627
  Male | 74 | 78 | 152
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 219 | 224 | 443
  Not Hispanic or Latino | 168 | 159 | 327
  Unknown or Not Reported | 2 | 7 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 15 | 22 | 37
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 141 | 134 | 275
  White | 46 | 58 | 104
  More than one race | 43 | 53 | 96
  Unknown or Not Reported | 138 | 117 | 255
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 389 | 390 | 779
Spoken Language [Count of Participants; unit: Participants] — Population: Participants were told to select their preferred language. Some participants declined to select one language.
  Participants
    English: number analyzed (Participants) | 372 | 371 | 743
    English | 292 | 290 | 582
    Spanish: number analyzed (Participants) | 372 | 371 | 743
    Spanish | 79 | 81 | 160
    Other: number analyzed (Participants) | 372 | 390 | 762
    Other | 1 | 0 | 1
Working Status [Count of Participants; unit: Participants]
  Unable to Work Due to Disability | 143 | 147 | 290
  Unemployed | 58 | 44 | 102
  Other | 188 | 199 | 387
Household Income Support [Count of Participants; unit: Participants] — Population: Row population differs from the overall because some participants declined to answer this question.
  Participants
    number analyzed (Participants) | 384 | 382 | 766
    No support | 114 | 103 | 217
    Any Support | 270 | 279 | 549
Participants Receiving Supplemental Security Insurance (SSI) [Count of Participants; unit: Participants]
  Not Receiving SSI | 212 | 173 | 385
  Receiving SSI | 177 | 217 | 394
Participants with Health Insurance Coverage [Count of Participants; unit: Participants]
  Medicaid | 301 | 288 | 589
  Private | 76 | 88 | 164
  None | 8 | 8 | 16
  Other | 4 | 6 | 10
Annual Household Income [Count of Participants; unit: Participants]
  Less than $20,000 | 183 | 179 | 362
  $20-$29,000 | 40 | 44 | 84
  $30-$39,000 | 41 | 30 | 71
  $40-$49,000 | 20 | 21 | 41
  Greater than $50,000 | 22 | 36 | 58
  Don't know / Refused | 83 | 80 | 163
Participants Reporting Opioid Use at baseline [Count of Participants; unit: Participants] — Population: Row population differs from the overall because some participants declined to answer this question.
  Participants
    number analyzed (Participants) | 381 | 384 | 765
    No | 275 | 291 | 566
    Yes | 106 | 93 | 199
Condition Participants were Referred to the Study for [Count of Participants; unit: Participants] — Each referring condition is not mutually exclusive. Participants were randomized based on their referring condition. Those who have multiple conditions are counted in the exclusive (back, neck, etc) categories and also in the multiple category.
  Participants
    Back pain | 261 | 273 | 534
    Neck pain | 70 | 68 | 138
    Osteoarthritis | 94 | 112 | 206
    Multiple conditions | 77 | 91 | 168
Depression Score as Measured by Patient Health Questionnaire 9 question (PHQ-9) Score [Mean (Standard Deviation); unit: Score on a scale] — The Patient Health Questionnaire 9 (PHQ9) consisting of 9 questions ranging from not at all (0 points) - nearly every day (3 points) and measures depression severity. The highest score is 27. A score 0-4 is considered minimal to none, 5-9 is mild, 10-14 is moderate, 15-19 is moderately severe, and 20-27 is severe.
  Score on a scale | 8.75 (6.02) | 8.74 (6.07) | 8.74 (6.04)
Patient Reported Global Health Score as Measured by The PROMIS-10 [Count of Participants; unit: Participants] — The Patient-Reported Outcomes Measurement Information System Global 10 (PROMIS-10) is a publically available questionnaire that allows for the measurement of quality of life for chronic conditions. It consists of 10 questions, scoring for the test can range from 8-40 (Raw score), the higher the score the worse the outcome. Those scores are changed into T scores that range from 32.4-85.2. The score is divided into categories. Physical health and mental health scores are calculated, which ranges from 4-20 (raw score each) each. Population: 1 participant in the individual arm declined to answer this question.
  Participants
    number analyzed (Participants) | 389 | 389 | 778
    Poor | 80 | 85 | 165
    Fair | 152 | 145 | 297
    Good | 111 | 104 | 215
    Very good | 33 | 42 | 75
    Excellent | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Pain Interference as Measured by the Brief Pain Inventory (BPI) (Intent to Treat Model)
Description: The Brief Pain Inventory (BPI) short form, is a self-reported questionnaire that serves as the primary measure of how much the participants' pain interferes with daily life. Pain interference is calculated using 7 questions that range from a score of 0 (no pain) to 10 (worst pain imaginable). The scores are added and divided by 7, therefore final scores can range from 0 - 10. Having a higher mean score indicates your pain severity is worse. Investigators measured improvement in BPI pain interference from baseline to week 24 (12 weeks after treatment window). The definition of intent to treat is all participants who were randomized into treatment. Statistical analysis only performed on baseline and week 12 (end of treatment) data.
Time Frame: Baseline, Week 12 (end of treatment window), and Week 24 (12 Weeks After Treatment Window)
Population: The data differs in participants from the overall data due to a few factors. Some participants did not complete the questionnaires for each time point. This may have been due to withdrawal, loss to follow up, or declining to answer a question. If a participant declined to answer a question their score could not be calculated which excludes them.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Group Acupuncture ITT: All the participants who were randomized to receive acupuncture weekly in a group acupuncture setting for 12 consecutive weeks.
- Individual Acupuncture ITT: All the participants who were randomized to receive acupuncture weekly in an individual acupuncture setting for 12 consecutive weeks.
Arm/Group | Group Acupuncture ITT | Individual Acupuncture ITT
Number analyzed (Participants) | 389 | 390
Units on a Scale
  Baseline: number analyzed (Participants) | 385 | 385
  Baseline | 6.0 (2.7) | 6.1 (2.7)
  Week 12: number analyzed (Participants) | 279 | 297
  Week 12 | 5.1 (3.0) | 4.8 (3.1)
  Week 24: number analyzed (Participants) | 266 | 277
  Week 24 | 5.3 (2.9) | 5.1 (3.1)
Statistical Analysis 1: Comparison: Group Acupuncture ITT vs Individual Acupuncture ITT; Test type: Superiority; p = 0.0691, ANCOVA; The outcome is the change of score from baseline to 12 weeks, adjusting for the baseline score; Mean Difference (Net) = -0.3714, 95% CI 2-sided [-0.7720 to 0.0291], Standard Error of Mean 0.2039 — The estimated value is the difference of score change from baseline to 12 weeks between two treatment arms (Individual-Group)

2. Primary Outcome: Pain Interference as Measured by the Brief Pain Inventory (BPI) (Per Protocol Model)
Description: The Brief Pain Inventory (BPI) short form, is a self-reported questionnaire that serves as the primary measure of how much your pain interferes with your life. Pain interference is calculated using 7 questions that range from a score of 0 (no pain) to 10 (worst pain imaginable). The scores are added and divided by 7, therefore final scores can range from 0 - 10. Having a higher mean score indicates your pain severity is worse. We measured improvement in BPI pain interference from baseline to week 24 (12 weeks after treatment window). The definition of Per Protocol is all participants who were randomized and who attended >=8 sessions of acupuncture. Statistical analysis only performed on baseline and week 12 (end of treatment) data.
Time Frame: Baseline, Week 12 (end of treatment window), and Week 24 (12 Weeks After Treatment Window))
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Group Acupuncture PP: All the participants who were randomized to receive acupuncture weekly in a group acupuncture setting for 12 consecutive weeks and attended >=8 sessions.
- Individual Acupuncture PP: All the participants who were randomized to receive acupuncture weekly in an individual acupuncture setting for 12 consecutive weeks and attended >=8 sessions.
Arm/Group | Group Acupuncture PP | Individual Acupuncture PP
Number analyzed (Participants) | 220 | 230
Units on a Scale
  Baseline: number analyzed (Participants) | 219 | 229
  Baseline | 5.8 (2.6) | 5.8 (2.8)
  Week 12: number analyzed (Participants) | 194 | 209
  Week 12 | 4.6 (2.9) | 4.5 (3.1)
  Week 24: number analyzed (Participants) | 180 | 189
  Week 24 | 5.1 (3.0) | 4.7 (3.1)
Statistical Analysis 1: Comparison: Group Acupuncture PP vs Individual Acupuncture PP; Test type: Superiority; p = 0.5077, ANCOVA; The outcome is the change of score from baseline to 12 weeks, adjusting for the baseline score; Mean Difference (Net) = -0.1631, 95% CI 2-sided [-0.6452 to 0.319], Standard Error of Mean 0.246 — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Improvement in Pain Interference as Measured by the Brief Pain Inventory (BPI) at Week 12 (Intent to Treat Model)
Description: The Brief Pain Inventory (BPI) short form, is a participant reported questionnaire that serves as the primary measure of how much your pain interferes with your life. It is a quality of life measure. Pain interference is calculated using 7 questions that range from a score of 0 (no pain) to 10 (worst pain imaginable). The scores are added and divided by 7, therefore final scores can range from 0 - 10. Having a higher score indicates your pain interference is worse. Respondent data is used for this analysis which shows whether participants experienced improvement in their pain interference from baseline to the end of treatment window (week 12). 30% improvement is a decrease of >=2 points on the BPI from baseline to the end of treatment window (week 12). A 30% decrease is considered a clinically significant improvement in pain. The definition of intent to treat is all participants who were randomized into treatment. Only participants who completed a week 12 questionnaire were analyzed.
Time Frame: Baseline, Week 12 (End of Treatment Window)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group Acupuncture ITT | Individual Acupuncture ITT
Number analyzed (Participants) | 271 | 288
Participants
  >=30% Improvement in Pain Interference | 82 | 108
  <30% Improvement in Pain Interference | 189 | 180
Statistical Analysis 1: Comparison: Group Acupuncture ITT vs Individual Acupuncture ITT; Test type: Non-Inferiority — The null hypothesis is that the group treatment is inferior to the individual treatment. 10% is set as the non-inferiority margin. If the upper limit of 90% confidence interval of the estimated value does not exceed 10%, non-inferiority is demonstrated; p = 0.24, Chi-squared; Risk Difference (RD) = 0.0724, 95% CI 2-sided [-0.0058 to 0.1506], Standard Error of Mean 0.0399 — The estimated value is the difference of proportion of respondents (>=30% improvement) at 12 weeks between two treatment arms (Individual-Group)

4. Primary Outcome: Improvement in Pain Interference as Measured by the Brief Pain Inventory (BPI) at Week 12 (Per Protocol Model)
Description: The Brief Pain Inventory (BPI) short form, is a self-reported questionnaire that serves as the primary measure of how much your pain interferes with your life. It is a quality of life measure. Pain interference is calculated using 7 questions that range from a score of 0 (no pain) to 10 (worst pain imaginable). The scores are added and divided by 7, therefore final scores can range from 0 - 10. Having a higher score indicates your pain interference is worse. Respondent data is used for this analysis which shows whether participants experienced improvement in pain interference from baseline to the end of treatment window (week 12). 30% improvement is a decrease of >=2 points on the BPI from baseline to the end of treatment window (week 12). A 30% decrease is considered a clinically significant improvement in pain. Per Protocol is all participants who were randomized and who attended >=8 sessions of acupuncture. Only participants who completed a week 12 questionnaire were analyzed.
Time Frame: Baseline, Week 12 (End of Treatment)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Group Acupuncture PP: All the participants who were randomized to receive acupuncture weekly in a group acupuncture setting for 12 consecutive weeks and attended >= 8 sessions.
- Individual Acupuncture PP: All the participants who were randomized to receive acupuncture weekly in an individual acupuncture setting for 12 consecutive weeks and attended >= 8 sessions.
Arm/Group | Group Acupuncture PP | Individual Acupuncture PP
Number analyzed (Participants) | 189 | 204
Participants
  >=30% Improvement in Pain Interference | 65 | 81
  <30% Improvement in Pain Interference | 124 | 123
Statistical Analysis 1: Comparison: Group Acupuncture PP vs Individual Acupuncture PP; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.17, Chi-squared; Risk Difference (RD) = 0.0531, 95% CI 2-sided [-0.0422 to 0.1485], Standard Error of Mean 0.0487 — [estimate comment as in outcome 3, analysis 1]

5. Primary Outcome: Improvement in Pain Interference as Measured by the Brief Pain Inventory (BPI) at Week 24 (Intent to Treat Model)
Description: The Brief Pain Inventory (BPI) short form, is a self-reported questionnaire that serves as the primary measure of how much your pain interferes with your life. It is a quality of life measure. Pain interference is calculated using 7 questions that range from a score of 0 (no pain) to 10 (worst pain imaginable). The scores are added and divided by 7, therefore final scores can range from 0 - 10. Having a higher score indicates your pain interference is worse. Respondent data is used for this analysis which shows whether participants experienced improvement in pain interference from baseline to week 24 (12 weeks after treatment window). 30% improvement is a decrease of >=2 points on the BPI from baseline to week 24 (12 weeks after treatment window). The definition of intent to treat is all participants who were randomized into treatment. Only participants who completed a week 24 questionnaire were included in the analysis.
Time Frame: Baseline, Week 24 (12 weeks after treatment window)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group Acupuncture ITT | Individual Acupuncture ITT
Number analyzed (Participants) | 268 | 283
Participants
  >=30% Improvement in Pain Interference | 77 | 99
  <30% Improvement in Pain Interference | 191 | 184
Statistical Analysis 1: Comparison: Group Acupuncture ITT vs Individual Acupuncture ITT; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.17, Chi-squared; Risk Difference (RD) = 0.0625, 95% CI 2-sided [-0.0151 to 0.1401], Standard Error of Mean 0.0396 — The estimated value is the difference of proportion of respondents (>=30% improvement) at 24 weeks between two treatment arms (Individual-Group)

6. Primary Outcome: Improvement in Pain Interference as Measured by the Brief Pain Inventory (BPI) at Week 24 (Per Protocol Model)
Description: The Brief Pain Inventory (BPI) short form, is a self-reported questionnaire that serves as the primary measure of how much your pain interferes with your life. It is a quality of life measure. Pain interference is calculated using 7 questions that range from a score of 0 (no pain) to 10 (worst pain imaginable). The scores are added and divided by 7, therefore final scores can range from 0 - 10. Having a higher score indicates your pain interference is worse. Respondent data is used for this analysis which shows whether participants experienced improvement in pain interference from baseline to week 24 (12 weeks after treatment). 30% improvement is a decrease of >=2 points on the BPI from baseline to week 24 (12 weeks after treatment). The definition of Per Protocol is all participants who have been randomized and who attended >=8 sessions of acupuncture. Only patients who completed a week 24 questionnaire were included in the analysis.
Time Frame: Baseline, Week 24 (12 weeks after treatment window)
Population: The data differs in participants from the overall data due to a few factors. Some participants did not complete the questionnaires for each time point. This may have been due to withdrawal, lost to follow up, or declining to answer a question. If a participant declined to answer a question their score could not be calculated which excludes them.
Measure: Count of Participants; unit: Participants
Arm/Group | Group Acupuncture PP | Individual Acupuncture PP
Number analyzed (Participants) | 182 | 197
Participants
  >=30% Improvement in Pain Interference | 56 | 78
  <30% Improvement in Pain Interference | 126 | 119
Statistical Analysis 1: Comparison: Group Acupuncture PP vs Individual Acupuncture PP; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.40, Chi-squared; Risk Difference (RD) = 0.0882, 95% CI 2-sided [-0.0075 to 0.184], Standard Error of Mean 0.0488 — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Pain Severity as Measured by the Brief Pain Inventory (BPI) (Intent to Treat Model)
Description: The Brief Pain Inventory (BPI) short form, is a self-reported questionnaire that serves as the measure of how severe your pain is. Pain severity is calculated using 4 questions that range from a score of 0 (no pain) to 10 (worst pain imaginable). The scores are added and then divided by 4, therefore final scores can range from 0 - 10. Having a higher mean score indicates your pain severity is worse. We measured improvement in BPI pain severity from baseline to week 24 (12 weeks after treatment window). The definition of intent to treat is anyone who intended to receive treatment; in our case, it is all participants who were randomized into treatment. Statistical analysis only performed on baseline and week 12 (end of treatment) data.
Time Frame: Baseline, Week 12 (end of treatment window), and Week 24 (12 Weeks After Treatment Window)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Group Acupuncture ITT | Individual Acupuncture ITT
Number analyzed (Participants) | 389 | 390
Units on a scale
  Baseline: number analyzed (Participants) | 389 | 386
  Baseline | 6.8 (1.8) | 6.8 (1.9)
  Week 12: number analyzed (Participants) | 285 | 301
  Week 12 | 5.7 (2.5) | 5.4 (2.7)
  Week 24: number analyzed (Participants) | 276 | 279
  Week 24 | 5.9 (2.6) | 5.8 (2.6)
Statistical Analysis 1: Comparison: Group Acupuncture ITT vs Individual Acupuncture ITT; Test type: Superiority; p = 0.1387, ANCOVA; The outcome is the change in score from baseline to 12 weeks, adjusting for the baseline score; Mean Difference (Net) = -0.2643, 95% CI 2-sided [-0.6136 to 0.0851], Standard Error of Mean 0.1782 — The estimated value is the difference of score change from baseline to 12 weeks between the two treatment arms (Individual-Group)

8. Secondary Outcome: Pain Severity as Measured by the Brief Pain Inventory (BPI) (Per Protocol Model)
Description: The Brief Pain Inventory (BPI) short form, is a self-reported questionnaire that serves as the measure of how severe your pain is. Pain severity is calculated using 4 questions that range from a score of 0 (no pain) to 10 (worst pain imaginable). The scores are added and divided by 4, therefore final scores can range from 0 - 10. Having a higher mean score indicates your pain severity is worse. We measured improvement in BPI pain severity from baseline to week 24 (12 weeks after treatment window). The definition of Per Protocol is all participants who were randomized and who attended >=8 sessions of acupuncture. Statistical analysis only performed on baseline and week 12 (end of treatment) data.
Time Frame: Baseline, Week 12 (end of treatment window), and Week 24 (12 Weeks After Treatment Window)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Group Acupuncture PP | Individual Acupuncture PP
Number analyzed (Participants) | 220 | 230
Units on a Scale
  Baseline: number analyzed (Participants) | 220 | 228
  Baseline | 6.7 (1.8) | 6.8 (1.9)
  Week 12: number analyzed (Participants) | 201 | 213
  Week 12 | 5.3 (2.4) | 5.1 (2.7)
  Week 24: number analyzed (Participants) | 190 | 191
  Week 24 | 5.7 (2.6) | 5.6 (2.5)
Statistical Analysis 1: Comparison: Group Acupuncture PP vs Individual Acupuncture PP; Test type: Superiority; p = 0.2725, ANCOVA; The outcome is the change in score from baseline to 12 weeks, adjusting for the baseline score; Mean Difference (Net) = -0.2334, 95% CI 2-sided [-0.6497 to 0.1829], Standard Error of Mean 0.2124 — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Improvement in Pain Severity as Measured by the Brief Pain Inventory (BPI) at Week 12 (Intent to Treat Model)
Description: The Brief Pain Inventory (BPI) short form, is a participant reported questionnaire that serves as the measure of how severe your pain is. Pain severity is calculated using 4 questions that range from a score of 0 (no pain) to 10 (worst pain imaginable). The scores are added and divided by 4, therefore final scores can range from 0 - 10. Having a higher mean score indicates your pain severity is worse. Respondent data is used for this analysis which shows whether participants experienced an improvement in their pain severity from baseline to the end of treatment window (week 12). 30% improvement is a decrease of >=2 points on the BPI from baseline to the end of treatment window (week 12). A 30% decrease in pain severity is considered a clinically significant improvement in pain. The definition of intent to treat is all participants who were randomized into treatment. Only participants who completed a week 12 questionnaire were analyzed.
Time Frame: Baseline, Week 12 (End of Treatment Window)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group Acupuncture ITT | Individual Acupuncture ITT
Number analyzed (Participants) | 285 | 299
Participants
  >=30% Improvement in Pain Severity | 87 | 104
  <30% Improvement in Pain Severity | 198 | 195
Statistical Analysis 1: Comparison: Group Acupuncture ITT vs Individual Acupuncture ITT; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.07, Chi-squared; Risk Difference (RD) = 0.0426, 95% CI 2-sided [-0.0334 to 0.1185], Standard Error of Mean 0.0388 — [estimate comment as in outcome 3, analysis 1]

10. Secondary Outcome: Improvement in Pain Severity as Measured by the Brief Pain Inventory (BPI) at Week 12 (Per Protocol Model)
Description: The Brief Pain Inventory (BPI) short form, is a participant reported questionnaire that serves as the measure of how severe your pain is. Pain severity is calculated using 4 questions that range from a score of 0 (no pain) to 10 (worst pain imaginable). The scores are added and divided by 4, therefore final scores can range from 0 - 10. Having a higher mean score indicates your pain severity is worse. Respondent data is used for this analysis which shows whether participants experienced an improvement in their pain severity from baseline to the end of treatment window (week 12). 30% improvement is a decrease of >=2 points on the BPI from baseline to the end of treatment window (week 12). A 30% decrease in pain severity is considered a clinically significant improvement in pain. The definition of Per Protocol is all participants who were randomized and who attended >=8 sessions of acupuncture. Only participants who completed a week 12 questionnaire were analyzed.
Time Frame: Baseline, Week 12 (End of Treatment Window)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group Acupuncture PP | Individual Acupuncture PP
Number analyzed (Participants) | 201 | 212
Participants
  >=30% Improvement in Pain Severity | 73 | 83
  <30% Improvement in Pain Severity | 128 | 129
Statistical Analysis 1: Comparison: Group Acupuncture PP vs Individual Acupuncture PP; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.07, Chi-squared; Risk Difference (RD) = 0.0283, 95% CI 2-sided [-0.0651 to 0.1218], Standard Error of Mean 0.0477 — [estimate comment as in outcome 3, analysis 1]

11. Secondary Outcome: Improvement in Pain Severity as Measured by the Brief Pain Inventory (BPI) at Week 24 (Intent to Treat Model)
Description: The Brief Pain Inventory (BPI) short form, is a participant reported questionnaire that serves as the measure of how severe your pain is. Pain severity is calculated using 4 questions that range from a score of 0 (no pain) to 10 (worst pain imaginable). The scores are added and divided by 4, therefore final scores can range from 0 - 10. Having a higher mean score indicates your pain severity is worse. Respondent data is used for this analysis which shows whether participants experienced an improvement in their pain severity from baseline to week 24 (12 weeks after treatment window). 30% improvement is a decrease of >=2 points on the BPI from baseline to week 24 (12 weeks after treatment window). A 30% decrease in pain severity is considered a clinically significant improvement in pain. The definition of intent to treat is all participants who were randomized into treatment. Only participants who completed a week 24 questionnaire were analyzed.
Time Frame: Baseline, Week 24 (12 Weeks After Treatment Window)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Group Acupuncture ITT | Individual Acupuncture ITT
Number analyzed (Participants) | 285 | 291
Participants
  >=30% Improvement in Pain Severity | 65 | 74
  <30% Improvement in Pain Severity | 220 | 217
Statistical Analysis 1: Comparison: Group Acupuncture ITT vs Individual Acupuncture ITT; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.02, Chi-squared; Risk Difference (RD) = 0.0262, 95% CI 2-sided [-0.0436 to 0.0961], Standard Error of Mean 0.0356 — [estimate comment as in outcome 5, analysis 1]

12. Secondary Outcome: Improvement in Pain Severity as Measured by the Brief Pain Inventory (BPI) at Week 24 (Per Protocol Model)
Description: The Brief Pain Inventory (BPI) short form, is a participant reported questionnaire that serves as the measure of how severe your pain is. Pain severity is calculated using 4 questions that range from a score of 0 (no pain) to 10 (worst pain imaginable). The scores are added and divided by 4, therefore final scores can range from 0 - 10. Having a higher mean score indicates your pain severity is worse. Respondent data is used for this analysis which shows whether participants experienced an improvement in their pain severity from baseline to week 24 (12 weeks after treatment window). 30% improvement is a decrease of >=2 points on the BPI from baseline to week 24 (12 weeks after treatment window). A 30% decrease in pain severity is considered a clinically significant improvement in pain. The definition of Per Protocol is all participants who have been randomized and who attended >=8 sessions of acupuncture. Only patients who completed a week 24 questionnaire were analyzed.
Time Frame: Baseline, Week 24 (12 Weeks After Treatment Window)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group Acupuncture PP | Individual Acupuncture PP
Number analyzed (Participants) | 196 | 202
Participants
  >=30% Improvement in Pain Severity | 48 | 56
  <30% Improvement in Pain Severity | 148 | 146
Statistical Analysis 1: Comparison: Group Acupuncture PP vs Individual Acupuncture PP; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.06, Chi-squared; Risk Difference (RD) = 0.0323, 95% CI 2-sided [-0.0539 to 0.1186], Standard Error of Mean 0.044 — [estimate comment as in outcome 5, analysis 1]

13. Secondary Outcome: Patient Global Impression of Change (PGIC) at Week 12 and Week 24 (Intent to Treat Model)
Description: The Patient Global Impression of Change (PGIC) is a self-reported questionnaire that indicates if a participant has perceived a change in their condition after having some sort of treatment. In this case, we evaluated whether the participants experienced a positive change after receiving treatment, a decrease in their pain, from baseline (before receiving treatment) to week 24 (12 weeks after treatment window). The PGIC is scored from 0 (much better) to 10 (much worse). A higher score indicates that a participant has felt worse since starting treatment. The definition of intent to treat is all participants who were randomized into treatment. Statistical analysis only performed on baseline and week 12 (end of treatment) data.
Time Frame: Week 12 (end of treatment window), and Week 24 (12 Weeks After Treatment Window)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Group Acupuncture ITT | Individual Acupuncture ITT
Number analyzed (Participants) | 389 | 390
Units on a Scale
  Week 12: number analyzed (Participants) | 295 | 310
  Week 12 | 3.0 (1.9) | 2.8 (1.9)
  Week 24: number analyzed (Participants) | 289 | 298
  Week 24 | 3.6 (2.3) | 3.3 (2.2)
Statistical Analysis 1: Comparison: Group Acupuncture ITT vs Individual Acupuncture ITT; Test type: Superiority; p = 0.1475, t-test, 2 sided; The outcome is the change of PGIC from baseline to 12 weeks; Mean Difference (Net) = -0.22, 95% CI 2-sided [-0.5288 to 0.0795], Standard Error of Mean 0.15 — The estimated value is the difference of PGIC change from baseline to 12 weeks between two treatment arms (Individual-Group)

14. Secondary Outcome: Patient Global Impression of Change (PGIC) at Week 12 and Week 24 (Per Protocol Model)
Description: The Patient Global Impression of Change (PGIC) is a self-reported questionnaire that indicates if a participant has perceived a change in their condition after having some sort of treatment. In this case, we evaluated whether the participants experienced a positive change after receiving treatment, a decrease in their pain, from baseline (before receiving treatment) to week 24 (12 weeks after treatment window). The PGIC is scored from 0 (much better) to 10 (much worse). A higher score indicates that a participant has felt worse since starting treatment. The definition of Per Protocol is all participants who were randomized and who attended >=8 sessions of acupuncture. Statistical analysis only performed on baseline and week 12 (end of treatment) data.
Time Frame: Week 12 (end of treatment window), and week 24 (12 weeks after treatment window)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Group Acupuncture PP | Individual Acupuncture PP
Number analyzed (Participants) | 220 | 230
Units on a Scale
  Week 12: number analyzed (Participants) | 207 | 220
  Week 12 | 2.6 (1.9) | 2.5 (1.9)
  Week 24: number analyzed (Participants) | 197 | 207
  Week 24 | 3.3 (2.3) | 3.0 (2.2)
Statistical Analysis 1: Comparison: Group Acupuncture PP vs Individual Acupuncture PP; Test type: Superiority; p = 0.3038, t-test, 2 sided; The outcome is the change of PGIC from baseline to 12 weeks; Mean Difference (Net) = -0.19, 95% CI 2-sided [-0.546 to 0.1706], Standard Error of Mean 0.18 — [estimate comment as in outcome 13, analysis 1]

15. Secondary Outcome: Improvement as Measured by the Patient Global Impression of Change (PGIC) at Week 12 (Intent to Treat Model)
Description: The Patient Global Impression of Change (PGIC) is a self-reported questionnaire that indicates if a patient has perceived a change in their condition after having some sort of treatment. Respondent data is used for this analysis which shows whether participants experienced improvement. Respondent data for the PGIC is scored using one question that ranges from 0 (no change or the condition got worse) to 7 (a great deal better). Improvement is defined as a score of >=6 points on the PGIC at week 12 (end of treatment window) as reported by the participants. The definition of intent to treat is all participants who were randomized into treatment. Only participants who completed a week 12 questionnaire were included in the analysis.
Time Frame: Week 12 (End of Treatment Window)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group Acupuncture ITT | Individual Acupuncture ITT
Number analyzed (Participants) | 294 | 309
Participants
  Improved (>=6 point score) | 103 | 116
  Not improved (<=5 point score) | 191 | 193
Statistical Analysis 1: Comparison: Group Acupuncture ITT vs Individual Acupuncture ITT; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.03, Chi-squared; Risk Difference (RD) = 0.0251, 95% CI 2-sided [-0.0517 to 0.1018], Standard Error of Mean 0.0392 — The estimated value is the difference of proportion of respondents (change post treatment>=6) at 12 weeks between two treatment arms (Individual-Group)

16. Secondary Outcome: Improvement as Measured by the Patient Global Impression of Change (PGIC) at Week 12 (Per Protocol Model)
Description: The Patient Global Impression of Change (PGIC) is a self-reported questionnaire that indicates if a patient has perceived a change in their condition after having some sort of treatment. Respondent data is used for this analysis which shows whether participants experienced improvement. Respondent data for the PGIC is scored using one question that ranges from 0 (no change or the condition got worse) to 7 (a great deal better). Improvement is defined as a score of >=6 points on the PGIC at week 12 (end of treatment window) as reported by the participants. The definition of Per Protocol is all participants who were randomized and who attended >=8 sessions of acupuncture. Only participants who completed a week 12 questionnaire were included in the analysis.
Time Frame: Week 12 (End of Treatment Window)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Individual Acupuncture ITT: All the participants who were randomized to receive acupuncture weekly in an individual acupuncture setting for 12 consecutive weeks and attended >=8 sessions.
Arm/Group | Group Acupuncture PP | Individual Acupuncture ITT
Number analyzed (Participants) | 206 | 219
Participants
  Improved (>=6 point score) | 89 | 95
  Not improved (<=5 point score) | 117 | 124
Statistical Analysis 1: Comparison: Group Acupuncture PP vs Individual Acupuncture ITT; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.02, Chi-squared; Risk Difference (RD) = 0.0018, 95% CI 2-sided [-0.0925 to 0.096], Standard Error of Mean 0.0481 — [estimate comment as in outcome 15, analysis 1]

17. Secondary Outcome: Improvement as Measured by the Patient Global Impression of Change (PGIC) at Week 24 (Intent to Treat Model)
Description: The Patient Global Impression of Change (PGIC) is a self-reported questionnaire that indicates if a patient has perceived a change in their condition after having some sort of treatment. Respondent data is used for this analysis which shows whether participants experienced improvement. Respondent data for the PGIC is scored using one question that ranges from 0 (no change or the condition got worse) to 7 (a great deal better). Improvement is defined as a score of >=6 points on the PGIC at week 24 (12 weeks after treatment window) as reported by the participants. The definition of intent to treat is all participants who were randomized into treatment. Only participants who completed a week 24 questionnaire were included in the analysis.
Time Frame: Week 24 (12 Weeks After Treatment Window
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group Acupuncture ITT | Individual Acupuncture ITT
Number analyzed (Participants) | 290 | 298
Participants
  Improved (>=6 point score) | 76 | 75
  Not improved (<=5 point score) | 214 | 223
Statistical Analysis 1: Comparison: Group Acupuncture ITT vs Individual Acupuncture ITT; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.00, Chi-squared; Risk Difference (RD) = -0.0104, 95% CI 2-sided [-0.081 to 0.0602], Standard Error of Mean 0.036 — The estimated value is the difference of proportion of respondents (change post treatment>=6) at 24 weeks between two treatment arms (Individual-Group)

18. Secondary Outcome: Improvement as Measured by the Patient Global Impression of Change (PGIC) at Week 24 (Per Protocol Model)
Description: The Patient Global Impression of Change (PGIC) is a self-reported questionnaire that indicates if a patient has perceived a change in their condition after having some sort of treatment. Respondent data is used for this analysis which shows whether participants experienced improvement. Respondent data for the PGIC is scored using one question that ranges from 0 (no change or the condition got worse) to 7 (a great deal better). Improvement is defined as a score of >=6 points on the PGIC at week 24 (12 weeks after treatment window) as reported by the participants. The definition of Per Protocol is all participants who were randomized and who attended >=8 sessions of acupuncture. Only participants who completed a week 24 questionnaire were included in the analysis.
Time Frame: Week 24 (12 Week After Treatment Window)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group Acupuncture PP | Individual Acupuncture ITT
Number analyzed (Participants) | 198 | 207
Participants
  Improved (>=6 point score) | 62 | 68
  Not improved (<=5 point score) | 136 | 139
Statistical Analysis 1: Comparison: Group Acupuncture PP vs Individual Acupuncture ITT; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.03, Chi-squared; Risk Difference (RD) = 0.0154, 95% CI 2-sided [-0.0755 to 0.1063], Standard Error of Mean 0.0464 — [estimate comment as in outcome 17, analysis 1]

19. Secondary Outcome: Participant Physical Health Score as Measured by the Patient-Reported Outcomes Measurement Information System 10 (PROMIS-10) (Intent to Treat Model)
Description: The Patient-Reported Outcomes Measurement Information System Global 10 (PROMIS-10) is a publically available questionnaire that allows for the measurement of quality of life for chronic conditions. It consists of 10 questions, for physical health only 4 questions are used, scoring for physical health can range from 4-20 (Raw score), the higher the score the better the outcome. The raw scores are changed into T-scores that range from 16.2-67.7. For this measure, we collected physical health scores from baseline to week 24 (12 weeks after treatment window). The definition of intent to treat is all participants who were randomized into treatment. Statistical analysis only performed on baseline and week 12 (end of treatment) data.
Time Frame: Baseline, Week 12 (end of treatment window), and Week 24 (12 Weeks After Treatment Window))
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Group Acupuncture ITT | Individual Acupuncture ITT
Number analyzed (Participants) | 389 | 390
T-score
  Baseline: number analyzed (Participants) | 385 | 387
  Baseline | 34.8 (7.2) | 34.8 (7.7)
  Week 12: number analyzed (Participants) | 295 | 308
  Week 12 | 38.5 (8.4) | 38.7 (8.3)
  Week 24: number analyzed (Participants) | 287 | 297
  Week 24 | 37.2 (8.7) | 37.8 (8.5)
Statistical Analysis 1: Comparison: Group Acupuncture ITT vs Individual Acupuncture ITT; Test type: Superiority; p = 0.8778, ANCOVA; The outcome is the change of score from baseline to 12 weeks, adjusting for the baseline score; Mean Difference (Net) = 0.082, 95% CI 2-sided [-0.9659 to 1.13], Standard Error of Mean 0.5336 — [estimate comment as in outcome 1, analysis 1]

20. Secondary Outcome: Participant Physical Health Score as Measured by the Patient-Reported Outcomes Measurement Information System 10 (PROMIS-10) (Per Protocol Model)
Description: The Patient-Reported Outcomes Measurement Information System Global 10 (PROMIS-10) is a publically available questionnaire that allows for the measurement of quality of life for chronic conditions. It consists of 10 questions, for physical health only 4 questions are used, scoring for physical health can range from 4-20 (Raw score), the higher the score the better the outcome. The raw scores are changed into T-scores that range from 16.2-67.7. For this measure, we collected physical health scores from baseline to week 24 (12 weeks after treatment window). The definition of Per Protocol is all participants who were randomized and who attended >=8 sessions of acupuncture. Statistical analysis only performed on baseline and week 12 (end of treatment) data..
Time Frame: Baseline, Week 12 (end of treatment window), and Week 24 (12 Weeks After Treatment Window)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Group Acupuncture PP | Individual Acupuncture PP
Number analyzed (Participants) | 220 | 230
T-score
  Baseline: number analyzed (Participants) | 217 | 228
  Baseline | 35.3 (7.1) | 35.2 (7.6)
  Week 12: number analyzed (Participants) | 207 | 219
  Week 12 | 39.4 (8.3) | 39.6 (8.1)
  Week 24: number analyzed (Participants) | 196 | 206
  Week 24 | 38.2 (8.7) | 38.7 (8.1)
Statistical Analysis 1: Comparison: Group Acupuncture PP vs Individual Acupuncture PP; Test type: Superiority; p = 0.5626, ANCOVA; The outcome is the change of score from baseline to 12 weeks, adjusting for the baseline score; Mean Difference (Net) = 0.3623, 95% CI 2-sided [-0.8667 to 1.5912], Standard Error of Mean 0.6252 — [estimate comment as in outcome 1, analysis 1]

21. Secondary Outcome: Improvement in Physical Health as Measured by Patient-Reported Outcomes Measure Information System 10 (PROMIS-10) at Week 12 (Intent to Treat Model)
Description: The Patient-Reported Outcomes Measurement Information System Global 10 (PROMIS-10) is a publically available questionnaire that allows for the measurement of quality of life for chronic conditions. The physical health score is calculated using 4 questions on the PROMIS-10 that range from 1 to 5. The score is then converted into a T score which can range from 16.2 to 67.7. The higher the score the better your physical health is. Improvement is categorized as an increase in the PROMIS-10 T-score from baseline to week 12 (end of treatment window), a >=2-point increase is considered a 30% improvement. The definition of intent to treat is all participants who have been randomized into treatment. Only patients who completed a week 12 questionnaire were included in the analysis.
Time Frame: Baseline, Week 12 (End of treatment window)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group Acupuncture ITT | Individual Acupuncture ITT
Number analyzed (Participants) | 291 | 306
Participants
  >=2 point Improvement in Physical health | 173 | 193
  <2 point Improvement in Physical health | 118 | 113
Statistical Analysis 1: Comparison: Group Acupuncture ITT vs Individual Acupuncture ITT; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.05, Chi-squared; Risk Difference (RD) = 0.0362, 95% CI 2-sided [-0.0419 to 0.1144], Standard Error of Mean 0.0399 — The estimated value is the difference of proportion of respondents (score change>=2) at 12 weeks between two treatment arms (Individual-Group)

22. Secondary Outcome: Improvement in Physical Health as Measured by Patient-Reported Outcomes Measure Information System 10 (PROMIS-10) at Week 12 (Per Protocol Model)
Description: The Patient-Reported Outcomes Measurement Information System Global 10 (PROMIS-10) is a publically available questionnaire that allows for the measurement of quality of life for chronic conditions. The physical health score is calculated using 4 questions on the PROMIS-10 that range from 1 to 5. The score is then converted into a T score which can range from 16.2 to 67.7. The higher the score the better your physical health is. Improvement is categorized as an increase in the PROMIS-10 T-score from baseline to week 12 (end of treatment window), a >=2-point increase is considered a 30% improvement. The definition of Per Protocol is all participants who have been randomized and who attended >=8 sessions of acupuncture. Only patients who completed a week 12 questionnaire were included in the analysis.
Time Frame: Baseline, Week 12 (End of Treatment Window)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group Acupuncture ITT | Individual Acupuncture ITT
Number analyzed (Participants) | 204 | 217
Participants
  >=2 point Improvement in Physical health | 125 | 147
  <2 point Improvement in Physical health | 79 | 70
Statistical Analysis 1: Comparison: Group Acupuncture ITT vs Individual Acupuncture ITT; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.22, Chi-squared; Risk Difference (RD) = 0.0647, 95% CI 2-sided [-0.0266 to 0.156], Standard Error of Mean 0.0466 — [estimate comment as in outcome 21, analysis 1]

23. Secondary Outcome: Improvement in Physical Health as Measured by Patient-Reported Outcomes Measure Information System 10 (PROMIS-10) at Week 24 (Intent to Treat Model)
Description: The Patient-Reported Outcomes Measurement Information System Global 10 (PROMIS-10) is a publically available questionnaire that allows for the measurement of quality of life for chronic conditions. The physical health score is calculated using 4 questions on the PROMIS-10 that range from 1 to 5. The score is then converted into a T score which can range from 16.2 to 67.7. The higher the score the better your physical health is. Improvement is categorized as an increase in the PROMIS-10 T-score from baseline to week 24 (12 weeks after treatment window), a >=2-point increase is considered a 30% improvement. The definition of intent to treat is all participants who were randomized into treatment. Only participants who completed a week 24 questionnaire were included in the analysis.
Time Frame: Baseline, Week 24 (12 Weeks After Treatment Window)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group Acupuncture ITT | Individual Acupuncture ITT
Number analyzed (Participants) | 283 | 296
Participants
  >=2 point Improvement in Physical health | 142 | 164
  <2 point Improvement in Physical health | 141 | 132
Statistical Analysis 1: Comparison: Group Acupuncture ITT vs Individual Acupuncture ITT; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.12, Chi-squared; Risk Difference (RD) = 0.0523, 95% CI 2-sided [-0.029 to 0.1335], Standard Error of Mean 0.0415 — The estimated value is the difference of proportion of respondents (score change>=2) at 24 weeks between two treatment arms (Individual-Group)

24. Secondary Outcome: Improvement in Physical Health as Measured by Patient-Reported Outcomes Measure Information System 10 (PROMIS-10) at Week 24 (Per Protocol Model)
Description: The Patient-Reported Outcomes Measurement Information System Global 10 (PROMIS-10) is a publically available questionnaire that allows for the measurement of quality of life for chronic conditions. The physical health score is calculated using 4 questions on the PROMIS-10 that range from 1 to 5. The score is then converted into a T score which can range from 16.2 to 67.7. The higher the score the better your physical health is. Improvement is categorized as a >= 2-point increase in the PROMIS-10 T-score from baseline to week 24 (12 weeks after treatment window). The definition of Per Protocol is all participants who were randomized and who attended >=8 sessions of acupuncture. Only participants who completed a week 24 questionnaire were included in the analysis.
Time Frame: Baseline, Week 24 (12 Weeks After Treatment Window)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group Acupuncture PP | Individual Acupuncture PP
Number analyzed (Participants) | 193 | 205
Participants
  >=2 point Improvement in Physical health | 96 | 121
  <2 point Improvement in Physical health | 97 | 84
Statistical Analysis 1: Comparison: Group Acupuncture PP vs Individual Acupuncture PP; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.44, Chi-squared; Risk Difference (RD) = 0.0928, 95% CI 2-sided [-0.0047 to 0.1903], Standard Error of Mean 0.0498 — [estimate comment as in outcome 23, analysis 1]

25. Secondary Outcome: Participant Mental Health Score as Measured by the Patient-Reported Outcomes Measurement Information System 10 (PROMIS-10) (Intent to Treat Model)
Description: The Patient-Reported Outcomes Measurement Information System Global 10 (PROMIS-10) is a publically available questionnaire that allows for the measurement of quality of life for chronic conditions. It consists of 10 questions, for mental health only 4 questions are used, scoring for mental health can range from 4-20 (Raw score), the higher the score the better the outcome. The raw scores are changed into T-scores that range from 21.2-67.6. For this measure, we collected mental health scores from baseline to week 24 (12 weeks after treatment window). The definition of intent to treat is all participants who were randomized into treatment. Statistical analysis only performed on baseline and week 12 (end of treatment) data.
Time Frame: Baseline, Week 12 (end of treatment window), and Week 24 (12 Weeks After Treatment Window)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Group Acupuncture ITT | Individual Acupuncture ITT
Number analyzed (Participants) | 389 | 390
T-score
  Baseline: number analyzed (Participants) | 385 | 384
  Baseline | 42.8 (9.8) | 42.4 (9.6)
  Week 12: number analyzed (Participants) | 291 | 308
  Week 12 | 43.8 (9.4) | 44.5 (9.6)
  Week 24: number analyzed (Participants) | 288 | 297
  Week 24 | 43.3 (9.9) | 44.1 (9.4)
Statistical Analysis 1: Comparison: Group Acupuncture ITT vs Individual Acupuncture ITT; Test type: Superiority; p = 0.4014, ANCOVA; The outcome is the change of score from baseline to 12 weeks, adjusting for the baseline score; Mean Difference (Net) = 0.4831, 95% CI 2-sided [-0.6468 to 1.6129], Standard Error of Mean 0.5753 — [estimate comment as in outcome 1, analysis 1]

26. Secondary Outcome: Participant Mental Health Score as Measured by the Patient-Reported Outcomes Measurement Information System 10 (PROMIS-10) (Per Protocol Model)
Description: The Patient-Reported Outcomes Measurement Information System Global 10 (PROMIS-10) is a publically available questionnaire that allows for the measurement of quality of life for chronic conditions. It consists of 10 questions, for mental health only 4 questions are used, scoring for mental health can range from 4-20 (Raw score), the higher the score the better the outcome. The raw scores are changed into T-scores that range from 21.2-67.6. For this measure, we collected mental health scores from baseline to week 24 (12 weeks after treatment window). The definition of Per Protocol is all participants who were randomized and who attended >=8 sessions of acupuncture. Statistical analysis only performed on baseline and week 12 (end of treatment) data.
Time Frame: Baseline, Week 12 (end of treatment window), and Week 24 (12 Weeks After Treatment Window)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Group Acupuncture PP | Individual Acupuncture PP
Number analyzed (Participants) | 220 | 230
T-Score
  Baseline: number analyzed (Participants) | 219 | 226
  Baseline | 43.6 (9.6) | 43.5 (9.7)
  Week 12: number analyzed (Participants) | 204 | 218
  Week 12 | 44.4 (9.2) | 45.2 (9.3)
  Week 24: number analyzed (Participants) | 198 | 206
  Week 24 | 44.1 (9.7) | 45.0 (9.0)
Statistical Analysis 1: Comparison: Group Acupuncture PP vs Individual Acupuncture PP; Test type: Superiority; p = 0.307, ANCOVA; The outcome is the change of score from baseline to 12 weeks, adjusting for the baseline score; Mean Difference (Net) = 0.6617, 95% CI 2-sided [-0.61 to 1.9334], Standard Error of Mean 0.647 — [estimate comment as in outcome 1, analysis 1]

27. Secondary Outcome: Improvement in Mental Health as Measured by Patient-Reported Outcomes Measure Information System 10 (PROMIS-10) at Week 12 (Intent to Treat Model)
Description: The Patient-Reported Outcomes Measurement Information System Global 10 (PROMIS-10) is a publically available questionnaire that allows for the measurement of quality of life for chronic conditions. The mental health score is calculated using 4 questions on the PROMIS-10 that range from 1 to 5. The score is then converted into a T score which can range from 21.2 to 67.6. The higher the score the better your mental health is. Improvement is categorized as an increase in the PROMIS-10 T-score from baseline to week 12 (end of treatment window), a >=5-point increase is what we used to measure improvement. The definition of intent to treat is all participants who were randomized into treatment. Only participants who completed a week 12 questionnaire were included in the analysis.
Time Frame: Baseline, Week 12 (End of Treatment Window)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group Acupuncture ITT | Individual Acupuncture ITT
Number analyzed (Participants) | 288 | 304
Participants
  >=5 point Improvement in Mental health | 75 | 84
  <5 point Improvement in Mental health | 213 | 220
Statistical Analysis 1: Comparison: Group Acupuncture ITT vs Individual Acupuncture ITT; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.01, Chi-squared; Risk Difference (RD) = 0.0159, 95% CI 2-sided [-0.0555 to 0.0873], Standard Error of Mean 0.0364 — The estimated value is the difference of proportion of respondents (score change>=5) at 12 weeks between two treatment arms (Individual-Group)

28. Secondary Outcome: Improvement in Mental Health as Measured by Patient-Reported Outcomes Measure Information System 10 (PROMIS-10) at Week 12 (Per Protocol Model)
Description: The Patient-Reported Outcomes Measurement Information System Global 10 (PROMIS-10) is a publically available questionnaire that allows for the measurement of quality of life for chronic conditions. The mental health score is calculated using 4 questions on the PROMIS-10 that range from 1 to 5. The score is then converted into a T score which can range from 21.2 to 67.6. The higher the score the better your mental health is. Improvement is categorized as an increase in the PROMIS-10 T-score from baseline to week 12 (end of treatment window), a >=5-point increase is what we used to measure improvement. The definition of Per Protocol is all participants who have been randomized and who attended >=8 sessions of acupuncture. Only patients who completed a week 12 questionnaire were included in the analysis.
Time Frame: Baseline, Week 12 (End of Treatment Window)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group Acupuncture PP | Individual Acupuncture PP
Number analyzed (Participants) | 203 | 215
Participants
  >=5 point Improvement in Mental health | 48 | 57
  <5 point Improvement in Mental health | 155 | 158
Statistical Analysis 1: Comparison: Group Acupuncture PP vs Individual Acupuncture PP; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.05, Chi-squared; Risk Difference (RD) = 0.0287, 95% CI 2-sided [-0.0544 to 0.1117], Standard Error of Mean 0.0424 — [estimate comment as in outcome 27, analysis 1]

29. Secondary Outcome: Improvement in Mental Health as Measured by Patient-Reported Outcomes Measure Information System 10 (PROMIS-10) at Week 24 (Intent to Treat Model)
Description: The Patient-Reported Outcomes Measurement Information System Global 10 (PROMIS-10) is a publically available questionnaire that allows for the measurement of quality of life for chronic conditions. The mental health score is calculated using 4 questions on the PROMIS-10 that range from 1 to 5. The score is then converted into a T-score which can range from 21.2 to 67.6. The higher the score the better your mental health is. Improvement is categorized as an increase in the PROMIS-10 T-score from baseline to week 24 (12 weeks after treatment window), a >=5-point increase is what we used to measure improvement. The definition of intent to treat is all participants who were randomized into treatment. Only participants who completed a week 24 questionnaire were included in the analysis.
Time Frame: Baseline, Week 24 (12 Weeks After Treatment Window)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group Acupuncture ITT | Individual Acupuncture ITT
Number analyzed (Participants) | 285 | 295
Participants
  >=5 point Improvement in Mental health | 72 | 86
  <5 point Improvement in Mental health | 213 | 209
Statistical Analysis 1: Comparison: Group Acupuncture ITT vs Individual Acupuncture ITT; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.05, Chi-squared; Risk Difference (RD) = 0.0389, 95% CI 2-sided [-0.0335 to 0.1112], Standard Error of Mean 0.0369 — The estimated value is the difference of proportion of respondents (score change>=5) at 24 weeks between two treatment arms (Individual-Group)

30. Secondary Outcome: Improvement in Mental Health as Measured by Patient-Reported Outcomes Measure Information System 10 (PROMIS-10) at Week 24 (Per Protocol Model)
Description: The Patient-Reported Outcomes Measurement Information System Global 10 (PROMIS-10) is a publically available questionnaire that allows for the measurement of quality of life for chronic conditions. The mental health score is calculated using 4 questions on the PROMIS-10 that range from 1 to 5. The score is then converted into a T-score which can range from 21.2 to 67.6. The higher the score the better your mental health is. Improvement is categorized as an increase in the PROMIS-10 T-score from baseline to week 24 (12 weeks after treatment window), a >=5-point increase is what we used to measure improvement. The definition of Per Protocol is all participants who were randomized and who attended >=8 sessions of acupuncture. Only participants who completed a week 24 questionnaire were included in the analysis.
Time Frame: Baseline, Week 24 (12 Weeks After Treatment Window)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group Acupuncture PP | Individual Acupuncture PP
Number analyzed (Participants) | 197 | 204
Participants
  >=5 point Improvement in Mental health | 45 | 59
  <5 point Improvement in Mental health | 152 | 145
Statistical Analysis 1: Comparison: Group Acupuncture PP vs Individual Acupuncture PP; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.18, Chi-squared; Risk Difference (RD) = 0.0608, 95% CI 2-sided [-0.0247 to 0.1463], Standard Error of Mean 0.0436 — [estimate comment as in outcome 29, analysis 1]

31. Secondary Outcome: Participants Who Reported Use of Prescription Opioids in the Last Week (Intent to Treat Model)
Description: Participants were asked whether they took any opioid medication within the last week. We compared self-reported prescription opioid use within a week of their baseline and week 12 questionnaires. The definition of intent to treat is all participants who have been randomized into treatment. Only participants who report having an opioid prescription are included in the analysis therefore if the participant did not have an opioid prescription they were excluded from the analysis. Statistical analysis only performed on baseline and week 12 (end of treatment) data.
Time Frame: Baseline, Week 12 (end of treatment window), and Week 24 (12 Weeks After Treatment Window)
Population: The data differs in participants from the overall data due to a few factors. Some participants did not complete the questionnaires for this time point. This may have been due to withdrawal, loss to follow up, or declining to answer this question. Only participants who responded to having taken prescription opioids were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Group Acupuncture ITT | Individual Acupuncture ITT
Number analyzed (Participants) | 389 | 390
Participants
  Opioid use within a week of Baseline: number analyzed (Participants) | 381 | 384
  Opioid use within a week of Baseline | 85 | 78
  Opioid use within a week of Week 12: number analyzed (Participants) | 290 | 306
  Opioid use within a week of Week 12 | 53 | 55
  Opioid use within a week of Week 24: number analyzed (Participants) | 285 | 291
  Opioid use within a week of Week 24 | 58 | 56
Statistical Analysis 1: Comparison: Group Acupuncture ITT vs Individual Acupuncture ITT; Two treatment arms are combined as one group to compare the outcome of interest pre- and post-randomization; Test type: Other — The null hypothesis is that there is no change in the proportion of participants with self-reported opioid prescription comparing 12 weeks vs baseline; p = 0.1658, McNemar

32. Secondary Outcome: Participants Who Reported Use of Prescription Opioids in the Last Week (Per Protocol Model)
Description: Participants were asked whether they took any opioid medication within the last week. We compared self-reported prescription opioid use within a week of their baseline and week 12 questionnaires. The definition of Per Protocol is all participants who have been randomized and who attended >=8 sessions of acupuncture. Only participants who report having an opioid prescription are included in the analysis therefore if the participant did not have an opioid prescription they were excluded from the analysis. Statistical analysis only performed on baseline and week 12 (end of treatment) data.
Time Frame: Baseline, Week 12 (end of treatment window), and Week 24 (12 Weeks After Treatment Window)
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Group Acupuncture PP | Individual Acupuncture PP
Number analyzed (Participants) | 220 | 230
Participants
  Opioid use within a week of Baseline: number analyzed (Participants) | 214 | 227
  Opioid use within a week of Baseline | 42 | 39
  Opioid use within a week of week 12: number analyzed (Participants) | 205 | 217
  Opioid use within a week of week 12 | 33 | 32
  Opioid use within a week of week 24: number analyzed (Participants) | 196 | 201
  Opioid use within a week of week 24 | 34 | 35
Statistical Analysis 1: Comparison: Group Acupuncture PP vs Individual Acupuncture PP; Two treatment arms are combined as one group to compare the outcome of interest pre- and post-randomization; Test type: Other — [test comment as in outcome 31, analysis 1]; p = 0.1172, McNemar

33. Secondary Outcome: Number of Days Participants Reported Using Prescription Opioids in the Last 7 Days (Intent to Treat Model)
Description: Participants were asked whether they took any opioid medication within the last week. If they did take any opioids in the last week we asked how many days they took their opioid medication. We collected data on the mean number of days participants took prescription opioid medication from baseline to week 24 (12 weeks after treatment window). The definition of intent to treat is all participants who were randomized into treatment. Statistical analysis only performed on baseline and week 12 (end of treatment) data.
Time Frame: Baseline, Week 12 (end of treatment window), and Week 24 (12 Weeks After Treatment Window)
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Days of Opioid use
Groups:
- Group Acupuncture ITT: All the participants who were randomized to receive acupuncture weekly in a group acupuncture setting for 12 consecutive weeks and had an active prescription for an opioid medication.
- Individual Acupuncture ITT: All the participants who were randomized to receive acupuncture weekly in an individual acupuncture setting for 12 consecutive weeks and had an active prescription for an opioid medication.
Arm/Group | Group Acupuncture ITT | Individual Acupuncture ITT
Number analyzed (Participants) | 389 | 390
Days of Opioid use
  Baseline: number analyzed (Participants) | 103 | 91
  Baseline | 4.3 (3.5) | 5.1 (2.8)
  12 weeks: number analyzed (Participants) | 65 | 66
  12 weeks | 4.2 (2.8) | 4.9 (3.6)
  24 weeks: number analyzed (Participants) | 72 | 65
  24 weeks | 4.5 (2.9) | 5.1 (2.8)
Statistical Analysis 1: Comparison: Group Acupuncture ITT vs Individual Acupuncture ITT; Two treatment arms are combined as one group to compare the outcome of interest prior- and post-randomization; Test type: Other — The null hypothesis is that there is no change in the days of self-reported opioid medication use comparing 12 weeks vs baseline; p = 0.0326, Wilcoxon signed rank test

34. Secondary Outcome: Number of Days Participants Reported Using Prescription Opioids in the Last 7 Days (Per Protocol Model)
Description: Participants were asked whether they took any opioid medication within the last week. If they did take any opioids in the last week we asked how many days they took their opioid medication. We collected data on the mean number of days participants took prescription opioid medication from baseline to week 24 (12 weeks after treatment window). The definition of Per Protocol is all participants who were randomized and who attended >=8 sessions of acupuncture. Statistical analysis only performed on baseline and week 12 (end of treatment) data.
Time Frame: Baseline, Week 12 (end of treatment window), and Week 24 (12 Weeks After Treatment Window)
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Days of Opioid use
Groups:
- Group Acupuncture PP: All the participants who were randomized to receive acupuncture weekly in a group acupuncture setting for 12 consecutive weeks, attended >=8 sessions and had an active prescription for an opioid medication.
- Individual Acupuncture PP: All the participants who were randomized to receive acupuncture weekly in an individual acupuncture setting for 12 consecutive weeks, attended >=8 sessions and had an active prescription for an opioid medication.
Arm/Group | Group Acupuncture PP | Individual Acupuncture PP
Number analyzed (Participants) | 220 | 230
Days of Opioid use
  Baseline: number analyzed (Participants) | 52 | 49
  Baseline | 4.0 (2.9) | 4.7 (3.0)
  12 weeks: number analyzed (Participants) | 41 | 42
  12 weeks | 3.6 (2.8) | 4.2 (3.2)
  24 weeks: number analyzed (Participants) | 44 | 41
  24 weeks | 4.1 (3.0) | 5.0 (2.9)
Statistical Analysis 1: Comparison: Group Acupuncture PP vs Individual Acupuncture PP; Two treatment arms are combined as one group to compare the outcome of interest prior- and post-randomization; Test type: Other — [test comment as in outcome 33, analysis 1]; p = 0.0026, Wilcoxon signed rank test

35. Secondary Outcome: Change in Participant Opioid Use in Milligrams of Morphine Equivalents (MME) Between 3 Months Pre and 3 Months Post-treatment Using Electronic Medical Record (EMR) Data (Intent to Treat Model)
Description: Milligrams of Morphine Equivalence (MME) is a value assigned to represent how strong an opioid is. It is determined by calculating a dose of morphine equivalent to the prescribed opioid. We compared the MME for participants who had Opioid prescriptions in their electronic medical records (EMR) during the 6 month period around treatment (3 months prior and post-treatment). A smaller MME indicates that the participant was using less medication. The definition of intent to treat is all participants who were randomized into treatment. The analysis is limited to participants who have documented opioid prescriptions in EMR. The change in MME was defined as post treatment minus pre treatment (in milligrams).
Time Frame: 6-Month Period Around Treatment Window (3 months pre- and 3 months post-treatment)
Population: The analysis is limited to participants who have documented opioid prescriptions in EMR. A participant could have a prescription in the pre-treatment period, post-treatment period or both.
Measure: Median (Inter-Quartile Range); unit: Milligrams of Morphine Equivalents
Groups:
- Group Acupuncture ITT: Participants who were randomized to receive acupuncture weekly in a group acupuncture setting for 12 consecutive week and had an active prescription for an opioid medication in EMR.
- Individual Acupuncture ITT: Participants who were randomized to receive acupuncture weekly in an individual acupuncture setting for 12 consecutive week and had an active prescription for an opioid medication in EMR.
Arm/Group | Group Acupuncture ITT | Individual Acupuncture ITT
Number analyzed (Participants) | 96 | 95
Milligrams of Morphine Equivalents | 0 [-3.0 to 8.8] | 0 [-12.8 to 3.0]
Statistical Analysis 1: Comparison: Group Acupuncture ITT vs Individual Acupuncture ITT; Test type: Superiority; p = 0.129, Wilcoxon (Mann-Whitney) — The change in MME was not normally distributed, thus we report median and IQR rather than mean/standard deviation. We employed Mann-Whitney to assess whether the change in MME between pre- and post-treatment periods differed across intervention arms

36. Secondary Outcome: Change in Participant Opioid Use in Milligrams of Morphine Equivalents (MME) Between 3 Months Pre and 3 Months Post-treatment Using Electronic Record (EMR) Data (Per Protocol Model)
Description: Milligrams of Morphine Equivalence (MME) is a value assigned to represent how strong an opioid is. It is determined by calculating a dose of morphine equivalent to the prescribed opioid. We compared the MME of participants who had Opioid prescriptions in their electronic medical records (EMR) during the 6 month period around treatment (3 months pre- and 3 months post-treatment). A smaller MME indicates that the participant was using less medication. The definition of Per Protocol is all participants who were randomized and who attended >=8 sessions of acupuncture. The analysis is limited to participants who have documented opioid prescriptions in EMR. The change in MME was defined as post treatment minus pre treatment (in milligrams).
Time Frame: 6-Month Period Around Treatment Window (3 months pre- and 3 months post-treatment)
Population: as for outcome 35
Measure: Median (Inter-Quartile Range); unit: Milligrams of Morphine Equivalents
Groups:
- Group Acupuncture PP: All the participants who were randomized to receive acupuncture weekly in a group acupuncture setting for 12 consecutive weeks, attended >=8 sessions and had an active prescription for an opioid medication in EMR (3 months pre- and 3 months post-treatment).
- Individual Acupuncture PP: All the participants who were randomized to receive acupuncture weekly in an individual acupuncture setting for 12 consecutive weeks, attended >=8 sessions and had an active prescription for an opioid medication in EMR around treatment (3 months pre- and 3 months post-treatment).
Arm/Group | Group Acupuncture PP | Individual Acupuncture PP
Number analyzed (Participants) | 46 | 53
Milligrams of Morphine Equivalents | 0 [-2.0 to 8.4] | -0.5 [-13.3 to 1.2]
Statistical Analysis 1: Comparison: Group Acupuncture PP vs Individual Acupuncture PP; Test type: Superiority; p = 0.031, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 35, analysis 1]

37. Secondary Outcome: Participants With Opioid Prescription Within a 6 Month Period Around Treatment Window According to Electronic Medical Record (EMR) Data (Intent to Treat Model)
Description: Participants' electronic medical records (EMR) were reviewed to see if they had a prescription for opioids during the 6-month period around their treatment window (3 months pre- and 3 months post-treatment). The definition of intent to treat is all participants who were randomized into treatment. There were 191 total participants that had "any documented opioid prescriptions in EMR.
Time Frame: 6-Month Period Around Treatment Window (3 months pre- and 3 months post-treatment)
Population: This analysis includes all participants who were randomized. A participant could have a prescription in the pre-treatment period, post-treatment period or both. Thus the total number of participants analyzed is not equal to the sum of participants in pre- and post-treatment periods.
Measure: Count of Participants; unit: Participants
Groups:
- Group Acupuncture ITT: Participants who were randomized to receive acupuncture weekly in a group acupuncture setting for 12 consecutive weeks and had an active prescription for an opioid medication in EMR.
- Individual Acupuncture ITT: Participants who were randomized to receive acupuncture weekly in an individual acupuncture setting for 12 consecutive weeks and had an active prescription for an opioid medication in EMR.
Arm/Group | Group Acupuncture ITT | Individual Acupuncture ITT
Number analyzed (Participants) | 389 | 390
Participants
  Opioid Prescription 3 Months Pre-Treatment | 51 | 64
  Opioid Prescription 3 Months Post-Treatment | 57 | 43
Statistical Analysis 1: Comparison: Group Acupuncture ITT vs Individual Acupuncture ITT; Test type: Superiority — Difference in change in proportion pre and post-treatment differs by treatment arm; p = 0.0059, Mixed Models Analysis

38. Secondary Outcome: Participants With Opioid Prescription Within a 6 Month Period Around Treatment Window According to Electronic Medical Record (EMR) Data ) (Per Protocol Model)
Description: Participants' electronic medical records (EMR) were reviewed to see if they had a prescription for opioids during the 6-month period around their treatment window (3 months pre- and 3 month post-treatment). The definition of Per Protocol is all participants who were randomized and who attended >=8 sessions of acupuncture.
Time Frame: 6-Month Period Around Treatment Window (3 months pre- and 3 months post-treatment)
Population: The analysis includes all participants who attended >= 8 sessions. A participant could have a prescription in the pre-treatment period, post-treatment period or both. Thus the total number of participants analyzed is not equal to the sum of participants in pre- and post-treatment periods.
Measure: Count of Participants; unit: Participants
Groups:
- Individual Acupuncture PP: All the participants who were randomized to receive acupuncture weekly in an individual acupuncture setting for 12 consecutive weeks, attended >=8 sessions and had an active prescription for an opioid medication in EMR (3 months pre- and 3 months post-treatment).
Arm/Group | Group Acupuncture PP | Individual Acupuncture PP
Number analyzed (Participants) | 220 | 230
Participants
  Opioid Prescription 3 Months Pre-Treatment | 26 | 35
  Opioid Prescription 3 Months Post-Treatment | 28 | 22
Statistical Analysis 1: Comparison: Group Acupuncture PP vs Individual Acupuncture PP; Test type: Superiority; p = 0.0385, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 24 weeks (12 weeks of treatment plus 12 weeks post-treatment)
Arm/Group | Group Acupuncture | Individual Acupuncture
All-Cause Mortality (participants affected / at risk) | 2/389 | 1/390
Serious Adverse Events (participants affected / at risk) | 0/389 | 0/390
Other Adverse Events (participants affected / at risk) | 10/389 | 5/390
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group Acupuncture (N=389) | Individual Acupuncture (N=390)
Prolonged Musculo-Skeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) — Procedural complication due to receiving acupuncture. Which may cause an increase in pain for some time.
Syncopal Symptoms (Nervous system disorders) | 4 (4) | 0 (0) — Procedural complication of receiving acupuncture because of the increased risk for fainting and lightheadedness.
Swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) — Procedural complication of receiving acupuncture. Swelling may occur.
Prolonged Bruising (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Bruising may be caused by acupuncture. It is also a side effect of Gua Sha.
Loss of vaccaria seed in ear (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Ear seed fell into the participant's ear. Seeds from the Vaccaria plant are secured on the ear with tape over acupuncture points. The seeds stimulate the point by exerting mild pressure. The patient can rub or press on them for an added effect.
Syncope (Nervous system disorders) | 1 (1) | 0 (0) — Participant fainted during treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT02456727/Prot_SAP_000.pdf